CLINICAL TRIAL: NCT06039423
Title: Modified Thoracoabdominal Nerves Block Through Perichondrial Approach: a New Strategy With a Wide Range of Utilization in Laparoscopic Gynecological Surgeries.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0306061
Record Dates: First submitted 2023-09-09; First posted 2023-09-15 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-07

CONDITIONS: Analgesic Efficacy of M-TAPA Block Accomplished Prior to Surgery in Patients Undergoing Laparoscopic Gynecological Surgeries
MeSH Terms: interventions — Ketorolac

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (M) (Active Comparator): The M-TAPA block will be combined with general anaesthesia.
  :
  Interventions: Procedure: The M-TAPA block
- Group (C) (Placebo Comparator): (control group) conventional general anaesthesia receiving multimodal analgesia.
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Procedure: The M-TAPA block — A high frequency (6-12 MHz) US linear probe was placed in the sagittal plane on the 10 th costal margin in the midline. The probe was then angulated deeply to visualize the lower surface of the costal cartilage. Via in plane technique, a 21 gauge Tuohy needle was inserted cranially between the lower fascia of the costal cartilage and upper fascia of the transversus abdominis muscle by moving the needle tip towards the posterior aspect of the 10 th costal cartilage and 20 mL bupivacaine (0.25 %) was injected.
  Arms: Group (M)
Drug: Ketorolac — conventional general anaesthesia receiving multimodal analgesia
  Arms: Group (C)

SUMMARY:
The current study was to assess the analgesic effects of the modified thoracoabdominal nerves block through perichondrial approach (M-TAPA) block in patients undergoing gynecological laparoscopic surgeries.The primary goal was to evaluate the analgesic efficacy of M-TAPA block accomplished prior to surgery in patients undergoing Laparoscopic gynecological surgeries

DETAILED DESCRIPTION:
All patients were thoroughly assessed preoperatively by history evaluation as regards current medical condition and drug therapy, careful clinical examination and laboratory evaluations (complete blood picture, liver function and renal function tests). Explanation of the anaesthesia method was done to all patients and they were instructed wisely on how to utilize the 10 cm linear visual Analogue scale (VAS), with (0) denoting pain free state, whereas (10) stands for the worst intractable pain [9]. Fifteen minutes before induction, all patients were premedicated with i.v. midazolam 0.03 mg kg-1 In the operating room, an i.v. cannula was placed and secured, then standard monitoring including (pulse oximetry, ECG, non- invasive blood pressure and end tidal carbon dioxide) were applied to each patient using multichannel (Datex ohmeda S/5, Germany) monitor. Anaesthesia was induced with lidocaine (1mg/kg) followed by (1.5 - 2 mg/kg) propofol -till cessation of verbal contact- and (1-1.5 μg/kg) fentanyl. Endotracheal intubation was accomplished with rocuronium (1mg/kg) and a suitable sized tube. Anaesthesia was maintained with sevoflurane (1-2 %) with (50 %) oxygen in air. Controlled mechanical ventilation was provided to maintain ETCO2 between (33-35 mmHg) and an oxygen saturation of 98 %.

Patients will be randomly assigned- using closed envelope technique- into 2 groups (30 patient) each:

Group (M): The M-TAPA block will be combined with general anaesthesia. Group (C): (control group) conventional general anaesthesia receiving multimodal analgesia.

In group (M), after the induction of anaesthesia and with the patient in the supine position, the block was performed before starting of the surgical procedure as described by Tulgar et al. [8]. After surgical skin disinfection with 10 % povidone-iodine, it was covered with sterile surgical fenestrated drapes. A high frequency (6-12 MHz) US linear probe (Fujifilm Sonosite, Tokyo, Japan) covered with a sterile cover was placed in the sagittal plane on the 10 th costal margin in the midline. The probe was then angulated deeply to visualize the lower surface of the costal cartilage. Via in plane technique, a 21 gauge Tuohy needle (Stimuplex B-Braun Medical, Melsungen, Germany) was inserted cranially between the lower fascia of the costal cartilage and upper fascia of the transversus abdominis muscle by moving the needle tip towards the posterior aspect of the 10 th costal cartilage with caution not to cross the cranial edge of the 10th costal cartilage and 20 mL of bupivacaine (0.25 %) was injected bilaterally, in the midclavicular line.

In group (C), ketorolac 0.75 mg/kg and paracetamol 10 mg/kg were administered intravenously before surgical stimulus.

Inadequate analgesia expressed in the form of elevated blood pressure or accelerated heart rate 20 % above baseline value was managed by administration of 0.5 (μg/kg) fentanyl bolus as a rescue analgesia. Perioperative hypothermia was managed by warming of i.v fluids and forced air warming to exposed areas. Precise fluid replacement was provided to all subjects according to the standard guidelines applied during anaesthesia.

At the end of surgery, sevoflurane vaporizer was shut off followed by administration of 100 % oxygen. Muscle relaxant was reversed with neostigmine 0.04 mg/kg and atropine 0.02 mg/kg slowly i.v, after oropharyngeal secretions were suctioned. The tube was removed after ensuring that the patients regained consciousness, breathed spontaneously and respond to verbal command. IV ondansetron (8) mg was given to all patients to guard against postoperative nausea and vomiting.

Patients were transferred to the PACU, where monitoring of heart rate, arterial blood pressure, respiration, and temperature were done by recovery nurses unaware to the study design to avoid bias. Postoperative analgesia was administrated with paracetamol i.v. 1 gm/8 hr throughout the first 24 hours postoperatively and standardized intravenous patient-controlled analgesia (IV-PCA) with morphine (0.5 mg/mL, 2-mg bolus, lock-out period 10 mins, and 4 hrs limit of 20 mg) based on reaching the score of ≥ (4) VAS.

ELIGIBILITY:
Inclusion Criteria:

* adult female patients
* aged 20-65 years,
* normal coagulation profile,
* scheduled for ambulatory laparoscopic gynecological surgeries under general anaesthesia.

Exclusion Criteria:

* patient refusal,
* skin infection at the site of the needle puncture
* known allergies to any of the study medications

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-07-02 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-09-07 (Actual)

PRIMARY OUTCOMES:
Total dose of fentanyl consumption | after 1 hour postoperative
  analgesic efficacy of M-TAPA block

SECONDARY OUTCOMES:
postoperative morphine given (mg) in the first 24 hrs | after 24 hours postoperatively
  analgesic efficacyof M-TAPA block

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria University Faculty of Medicin, Alexandria, Egypt